CLINICAL TRIAL: NCT06143995
Title: The Diagnosis and Treatment Pattern of CKD in Patients With Cardiovascular Disease- a National Cross-sectional Study
Acronym: CREATIVE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY2023-267-01
Record Dates: First submitted 2023-08-20; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-07

CONDITIONS: Renal Insufficiency, Chronic; Cardiovascular Diseases; Diagnosis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about in a total of approximately 2000 patients with cardiovascular disease recruited from about 25 participating sites in China with eGFR<60 ml/min/1.73 m2 and/or UACR>30 mg/g at least twice 3 months apart within the previous 12 months who had been hospitalized in the cardiology department within the previous 12 months. The main questions it aims to answer are:

* To estimate the diagnosis rate of CKD in patients with cardiovascular disease and laboratory evidence of CKD
* To describe the CKD awareness and treatment pattern in patients with cardiovascular disease and laboratory evidence of CKD.
* To describe the socio-demographic and clinical characteristics of CKD in patients with cardiovascular disease and laboratory evidence of CKD

Participants will be invited to undergo a baseline visit, and the demographics, lifestyle factors, clinical characteristics, and laboratory tests will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Female and/or male aged ≥18 years
2. Admitted to the cardiology department with diagnosed cardiovascular disease within the previous 12 months
3. Participants with eGFR<60 ml/min/1.73 m2 and/or UACR>30 mg/g at least twice 3 months apart within the previous 12 months

Exclusion Criteria:

1. Participants with known eGFR<20 ml/min/1.73 m2 or undergoing dialysis or kidney transplantation
2. Pregnant or lactating women
3. Exposure to contrast medium or other reason leading to potential acute kidney injury since the baseline examination of eGFR/UACR
4. Patients who were participating in or had participated in any other clinical trial within the previous 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: a total of approximately 2000 patients with cardiovascular disease recruited from about 25 participating sites in China
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
CKD diagnosis rates | 1 day
  CKD diagnosis rates in overall enrolled patients and subgroups (stratified by isolated estimated glomerular filtration rate (eGFR) measurement, isolated urinary albumin-to-creatinine ratio ( UACR) measurement, and both measurements) will be assessed in 12 month.

SECONDARY OUTCOMES:
Clinical characteristics | 1 day
  Clinical characteristics in the overall participants and groups stratified by CKD diagnosis (CKD diagnosis, and CKD non-diagnosis) will be reported in 12 months.
CKD diagnosis/treatment rate | 1 day
  CKD diagnosis/treatment rate in groups stratified by of disease types (HTN, Coronary artery disease (CAD), Heart Failure (HF), type 2 diabetes mellitus (T2DM), etc.) will be assessed in 12 months.
The number, types, treatment rates of medicine | 1 day
  The number, types, treatment rates of medicine (by class) for renal protection or with potential renal contraindication, awareness in the overall enrolled participants and groups stratified by CKD diagnosis (CKD diagnosis, CKD non-diagnosis) will be reported in 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China